CLINICAL TRIAL: NCT06543043
Title: An Open-Label, Parallel Group Study Designed to Investigate the Effect of the CYP3A Inducer Phenytoin and the CYP3A Inhibitor Itraconazole on the Pharmacokinetics of Sonrotoclax (BGB-11417) in Healthy Subjects
Brief Title: A Study to Evaluate the Effects of Phenytoin and Itraconazole on Sonrotoclax (BGB-11417) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BGB-11417-107; QSC302214 (Other: Quotient Sciences)
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Not Determined
Keywords: sonrotoclax; BGB-11417; healthy volunteers; phenytoin; itraconazole
MeSH Terms: interventions — Phenytoin; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Phenytoin + Sonrotoclax (Experimental): Part A is designed to determine the effect of multiple doses of phenytoin on sonrotoclax in healthy participants.
  Interventions: Drug: Phenytoin; Drug: sonrotoclax
- Part B: Itraconazole + Sonrotoclax (Experimental): Part B is designed to determine the effect of multiple doses of itraconazole on sonrotoclax in healthy participants.
  Interventions: Drug: Itraconazole; Drug: sonrotoclax

INTERVENTIONS:
Drug: Phenytoin — Administered orally.
  Arms: Part A: Phenytoin + Sonrotoclax
Drug: Itraconazole — Administered orally.
  Arms: Part B: Itraconazole + Sonrotoclax
Drug: sonrotoclax — Administered orally.
  Other Names: BGB-11417

SUMMARY:
This is a single-center, open-label, parallel group study designed to investigate the effect of CYP3A induction and inhibition following multiple doses of phenytoin (Part A) and itraconazole (Part B), respectively, on the pharmacokinetics of sonrotoclax in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign a written informed consent
* Able and willing to comply with all study requirements
* Healthy males or healthy females of non-childbearing potential
* Agrees to use an adequate method of contraception
* Body mass index (BMI) of 18.0 to 32.0 kg/m^2 as measured at screening or, if outside the range, considered not clinically significant by the investigator.

Exclusion Criteria:

* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency (HIV) antibody results
* Prior treatment with sonrotoclax
* Evidence of renal impairment at screening
* Any contraindication to the use of phenytoin (Part A) or itraconazole (Part B)
* Current smokers and those who have smoked within the last 12 months
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* History of any drug or alcohol abuse in the past 2 years
* Serious adverse reaction or serious hypersensitivity to any drug or formulation excipients
* History of clinically significant disorders as judged by the investigator

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Parts A and B: Lag time before observation of quantifiable concentrations in plasma (Tlag) of sonrotoclax | Approximately 21 days for Part A and 11 days for Part B
Parts A and B: Time to maximum observed concentration (Tmax) of sonrotoclax | Approximately 21 days for Part A and 11 days for Part B
Parts A and B: Maximum observed plasma concentration (Cmax) of sonrotoclax | Approximately 21 days for Part A and 11 days for Part B
Parts A and B: Area under the concentration time curve from time zero up to the last quantifiable concentration (AUClast) of sonrotoclax | Approximately 21 days for Part A and 11 days for Part B
Parts A and B: Area under the concentration time curve from time zero extrapolated to infinity (AUCinf) of sonrotoclax | Approximately 21 days for Part A and 11 days for Part B
Parts A and B: Terminal phase elimination rate constant (lambda-z) of sonrotoclax | Approximately 21 days for Part A and 11 days for Part B
Parts A and B: Terminal elimination half life (T1/2) of sonrotoclax | Approximately 21 days for Part A and 11 days for Part B
Parts A and B: Apparent oral clearance (CL/F) of sonrotoclax | Approximately 21 days for Part A and 11 days for Part B
Parts A and B: Apparent volume of distribution (Vz/F) of sonrotoclax | Approximately 21 days for Part A and 11 days for Part B

SECONDARY OUTCOMES:
Parts A and B: Number of Participants with Adverse Events (AEs) | From time of providing written informed consent until up to 30 days after the final dose of study treatment for each part of the study; approximately 8 weeks for Part A and approximately 7 weeks for Part B
  Number of participants with AEs and SAEs, including findings from vital signs, electrocardiograms (ECGs), physical examinations, and clinical laboratory assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (1):
- Quotient Sciences, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes